CLINICAL TRIAL: NCT00796380
Title: Clinical Study of Xingnaojing for the Treatment of Convulsive Diseases
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shenzhen Children's Hospital (Other Government)
Responsible Party: Epilepsy and cerebral palsy center, Shenzhen Children's Hospital, Shenzhen Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ChiCTR-TNC-00000097
Record Dates: First submitted 2008-11-21; First posted 2008-11-24 (Estimated); Last update posted 2008-11-24 (Estimated); Status verified 2008-11

CONDITIONS: Convulsive Diseases
MeSH Terms: interventions — xingnaojing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Xingnaojing — injection

SUMMARY:
The purpose of this study is to evaluate the efficacy of Xingnaojing for the treatment of convulsive diseases; to investigate whether convulsion episodes can be induced or aggravated by Xingnaojing and the role inflammation plays in the process.

ELIGIBILITY:
Inclusion Criteria:

1. Febrile convulsion: positive family history of febrile convulsion; aged between 6 months and 6 years old; in accordance with the diagnosis criteria of simple type of febrile convulsion
2. Frequent episodes of epilepsy: epilepsy episodes of all types; > 3 times / week
3. Refractory epilepsy: no satisfactory efficacy after treatment by 2~3 antiepileptic drugs; ≥ 1 time / month
4. Cerebral palsy: all types of cerebral palsy in children less than 3 years old. -

Exclusion Criteria:

1. Febrile convulsion: family history of epilepsy, complex type of febrile convulsion, epileptic episodes, febrile convulsion plus
2. Frequent episodes of epilepsy: combined with advanced diseases
3. Refractory epilepsy: epilepsy combined with advanced diseases
4. Cerebral palsy: advanced diseases combined with backwardness or retardation of brain function development.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-11 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Antipyretic rate , Frequency of convulsive episodes , | one year
Frequency of convulsive episodes | 1 year